CLINICAL TRIAL: NCT01441167
Title: VRC 312: A Phase 1, Open-Label, Dose-Escalation Clinical Trial With Experimental Challenge to Evaluate Intravenous Administration of the PfSPZ Vaccine in Malaria-Naive Adults
Brief Title: Experimental PfSPZ Vaccine in Adults Without Malaria
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: Sanaria Incorporated (Unknown); U.S. Military Malaria Vaccine Program (Unknown)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 110257; 11-I-0257
Record Dates: First submitted 2011-09-24; First posted 2011-09-27 (Estimated); Last update posted 2018-07-05 (Actual); Status verified 2013-06-05

CONDITIONS: Malaria; Prevention and Control; Acquired Immunity
Keywords: Healthy Subjects; Immunogenicity; Vaccine-Mediated Protection; Sporozoites; Parasitemia; Healthy Volunteer; HV
MeSH Terms: conditions — Malaria; Parasitemia

INTERVENTIONS:
Biological: PfSPZ

SUMMARY:
Background:

* Malaria parasites are carried by mosquitoes, which spread the infection by biting people. Currently, there is no effective malaria vaccine. However, studies show that volunteers bitten many times by mosquitoes that carry weakened malaria parasites could fight off getting sick with malaria when later exposed to normal malaria parasites. Malaria parasites are weakened by exposing them to radiation when they are in the stage of development called sporozoites . Only the mosquitoes are irradiated and study volunteers are not exposed to radiation. The radiation stops the parasites from being able to cause disease but still promote protection. For many years, it was not possible to give these sporozoites to people as a vaccine since they could not be adequately purified from the mosquito. Scientists have recently figured out how to produce and isolate the weakened sporozoites so that they can be given in an injected vaccine. This vaccine is known as the "PfSPZ vaccine".
* A malaria challenge will be used to test whether the vaccine will prevent infection. In a malaria challenge, mosquitoes that have the malaria parasite will be allowed to bite a participant's arm. In the event that the vaccine does not work, the malaria parasite used for the challenge can be treated completely with common anti-malaria medications. Participants will be treated immediately if they develop malaria symptoms.

Objectives:

- To test the safety and effectiveness of the PfSPZ vaccine.

Eligibility:

- Healthy volunteers between 18 to 45 years of age.

Design:

* Participants will be screened with a physical exam, medical history, and blood tests. There will be five different groups of study participants, all of whom will be monitored with frequent blood tests.
* Group 1 will have two vaccines with the lowest amount of the vaccine given 4 weeks apart, with regular clinic visits up to 24 weeks after the second vaccine. This group will not have a malaria challenge.
* Group 2 will have four or six vaccines given 4 weeks apart at a higher dose than group 1. A malaria challenge will be given about 3 weeks after the last vaccine. Follow-up visits will continue through 24 weeks after the last vaccine.
* Group 3 will have four or six vaccines given 4 weeks apart at a higher dose than group 2. A malaria challenge will be given about 3 weeks after the last vaccination, as for Group 2. Follow-up visits will continue through 24 weeks after last vaccine.
* Group 4 will have four or six vaccines given 4 weeks apart at a higher dose than group 3. A malaria challenge will be given about 3 weeks after the last vaccination. Follow up visits will continue through 24 weeks after last vaccine.
* Group 5 will serve as a control group and will not receive the vaccine, but will have the malaria challenge. Follow-up visits will continue through 8 weeks after the challenge.

All participants from any group who receive a malaria challenge will be treated promptly for malaria when it develops.

DETAILED DESCRIPTION:
Study Design: VRC 312 is the second study of the PfSPZ Vaccine and the first study to evaluate intravenous (IV) administration of this vaccine. The study is designed as an openlabel evaluation of the safety, tolerability, immunogenicity and protective efficacy of the vaccine at successively higher dosages (2000; 7500; 30,000 and 135,000 SPZ per injection) administered by the IV route. The 3 higher dosages will be evaluated for protection against a malaria challenge after 4 to 6 vaccinations. Control subjects are included in the malaria challenge. The primary objectives of the study are related to the safety and tolerability of the vaccine at the 4 dosage levels when administered IV; the secondary objectives are related to PfSPZ vaccine-mediated protection against Plasmodium falciparum (Pf) challenge at the 3 higher dosage levels; and the exploratory objectives are related to the immunogenicity of the PfSPZ Vaccine and defining an immune correlate of protection.

Product Description: The investigational PfSPZ Vaccine is manufactured by Sanaria, Inc (Rockville, MD) under current Good Manufacturing Practices (cGMP). The vaccine consists of a suspension of purified, metabolically-active, radiation-attenuated cryopreserved Pf sporozoites formulated in cryoprotectant and dispensed in a 0.5 mL screw-cap vial containing a 20 mcL aliquot at a concentration of 150,000 sporozoites (+/-50,000 sporozoites) per 20 mcL. The vaccine is stored in the vapor-phase of liquid nitrogen (LNVP) at -140 to -196 degrees C. The PfSPZ Vaccine is delivered by Sanaria, Inc. to the clinical investigators and diluted in phosphate buffered saline (PBS) with 1% human serum albumin (HSA) to achieve the correct dosage.

Subjects: Healthy subjects, 18-45 years old, who are malaria-naive. The fewest number of subjects needed to complete the study as originally designed was 51; however, with inclusion of study provisions for back-up challenge subjects enrollment of additional vaccinees and options for rechallenge, as added by protocol amendments, the amended accrual allowance is 68 subjects.

Study Plan: Subjects will be enrolled in a step-wise, dose-escalation manner with stringent stopping rules designed for subject safety. The first 12 subjects will be allocated as the pilot subjects that comprise Groups 1, 2a, 3a, 4a; each of which includes 3 pilot subjects. For the pilot subjects, the 1st vaccination (V1) and 2nd vaccination (V2) will be administered no faster than one per pilot subject every 2 hours.

Before administration of the first dose to the subsequent pilot Group (dose escalation), at least 5 weeks of cumulative safety data for the pilot subjects in a dosage group (i.e., 1 week past 2nd vaccination) must be submitted to the Safety Monitoring Committee (SMC) and the FDA, and protocol-specified approval received for the dose escalation.

Subjects in vaccine Groups 2, 3, 4 and the Group 5 controls will be challenged by exposure to Anopheles stephensi mosquitoes infected with Pf sporozoites in a controlled setting, followed by testing for parasitemia at specified intervals through up to 28 days post-challenge. To facilitate intensive daily close monitoring of clinical status and blood smears, 11 overnight stays are required from days 7-18 post-challenge. Subjects who develop blood stage P. falciparum infection will be treated as soon as a case is identified by the protocol criteria. Following treatment, a subject will be considered cured when 2 consecutive daily blood smears are negative. After establishing cure, blood smear checks may end and the subject may discontinue overnight stays.

Challenges occur at specified timepoints in which each challenge includes vaccine recipients and control subjects. Rechallenge options to assess for durability of protective responses and further evaluation of immune correlates of protection are included in the protocol.

Study Duration: The study will take approximately 18 months to complete. The period of follow-up for each vaccinated subject is through at least 24 weeks after the last vaccination. The total duration on study will vary depending upon the schedule assignment and whether or not the subject participates in a rechallenge. The Group 5 (challenge only) subjects and rechallenged subjects will be followed through 8 weeks after last challenge.

ELIGIBILITY:
* INCLUSION CRITERIA:

A volunteer must meet all of the following criteria to be included:

1. 18 to 45 years old adults.
2. Able and willing to participate for the duration of the study.
3. Able to provide proof of identity to the satisfaction of the study clinician completing the enrollment process.
4. Able and willing to complete the informed consent process.
5. Willing to donate blood for sample storage to be used for future research.
6. Willing to refrain from blood donation to blood banks for 3 years following P. falciparum challenge.
7. Agree not to travel to a malaria endemic region during the entire course of study participation.
8. Physical examination and laboratory results without clinically significant findings and a body mass index (BMI) less than or equal to 35 for Groups 1, 2, 3 and 4 or BMI less than or equal to 40 for Group 5.

   LABORATORY CRITERIA WITHIN 56 DAYS PRIOR TO ENROLLMENT:
9. Hemoglobin greater than or equal to 11.2 g/dL for women; greater than or equal to 13.0 g/dL for men.
10. Differential and platelet count either within institutional normal range or accompanied by site physician approval.
11. Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) less than or equal to 1.25 times upper limit of normal (ULN) for Groups 1, 2, 3 and 4 or less than or equal to 1.75 ULN for Group 5.
12. Serum creatinine less than or equal to upper limit of normal.
13. Negative for HIV infection.

    LABORATORY CRITERION DOCUMENTED ANY TIME PRIOR TO ENROLLMENT:
14. Negative sickle cell screening test.

    FEMALE-SPECIFIC CRITERIA:
15. Negative beta-HCG pregnancy test (urine or serum) on day of enrollment for women presumed to be of childbearing potential.
16. A woman of childbearing potential must agree to use an effective means of birth control throughout the duration of study participation.

EXCLUSION CRITERIA:

A volunteer will be excluded if one or more of the following conditions apply:

1. Woman who is breast-feeding or planning to become pregnant during the time interval needed to complete the study.
2. Receipt of a malaria vaccine in a prior clinical trial.
3. Any history of malaria infection.
4. Evidence of increased cardiovascular disease risk; defined as >10% five year risk by the non-laboratory method.
5. Screening EKG showing pathologic Q waves and significant ST-T wave changes; left ventricular hypertrophy; any non-sinus rhythm (except isolated premature atrial contractions); left bundle branch block; or advanced (secondary or tertiary) A-V heart block.
6. Current use of systemic immunosuppressant pharmacotherapy.
7. History of a splenectomy, sickle cell disease or sickle cell trait.
8. Plan for major surgery between enrollment and challenge.
9. Known allergy to any component of the vaccine formulation; history of anaphylactic response to mosquito-bites; or known allergy to chloroquine phosphate, atovaquone or proguanil.
10. Participation in any study involving another investigational vaccine or drug within 12 weeks prior to enrollment, or plan to participate in another investigational vaccine/drug research during the study.
11. Personal beliefs that prohibit the receiving of vaccine product containing human serum albumin within the diluent.
12. Use or planned use of any drug with anti-malarial activity that would coincide with study vaccination or challenge.
13. History of psoriasis or porphyria, which may be exacerbated after treatment with chloroquine.
14. Anticipated use of medications known to cause drug reactions with chloroquine or atovaquone-proguanil (Malarone) such as cimetidine, metoclopramide, antacids, and kaolin.
15. Psychiatric condition that precludes compliance with the protocol; past or present psychoses; disorder requiring lithium; or within five years prior to enrollment, history of a suicide plan or attempt.
16. Any medical, psychiatric, social condition, occupational reason or other responsibility that, in the judgment of the investigator, is a contraindication to protocol participation or impairs a volunteer s ability to give informed consent.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 64 (Actual)
Dates: Start 2011-09-14; Primary Completion 2013-06-05 (Actual); Study Completion 2013-06-05 (Actual)

PRIMARY OUTCOMES:
The primary objectives of the study are related to the safety and tolerability of the vaccine at the 4 dosage levels when administered IV.

SECONDARY OUTCOMES:
The secondary objectives are related to PfSPZ vaccine-mediated protection against Plasmodium falciparum (Pf) challenge at the 3 higher dosage levels.

CONTACTS AND LOCATIONS:
Overall Officials: Robert A Seder, M.D., Principal Investigator — National Institute of Allergy and Infectious Diseases (NIAID)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Sachs J, Malaney P. The economic and social burden of malaria. Nature. 2002 Feb 7;415(6872):680-5. doi: 10.1038/415680a. PMID 11832956
- [Background] Breman JG. Eradicating malaria. Sci Prog. 2009;92(Pt 1):1-38. doi: 10.3184/003685009X440290. PMID 19544698
- [Background] Nussenzweig RS, Vanderberg J, Most H, Orton C. Protective immunity produced by the injection of x-irradiated sporozoites of plasmodium berghei. Nature. 1967 Oct 14;216(5111):160-2. doi: 10.1038/216160a0. No abstract available. PMID 6057225
- [Derived] Seder RA, Chang LJ, Enama ME, Zephir KL, Sarwar UN, Gordon IJ, Holman LA, James ER, Billingsley PF, Gunasekera A, Richman A, Chakravarty S, Manoj A, Velmurugan S, Li M, Ruben AJ, Li T, Eappen AG, Stafford RE, Plummer SH, Hendel CS, Novik L, Costner PJ, Mendoza FH, Saunders JG, Nason MC, Richardson JH, Murphy J, Davidson SA, Richie TL, Sedegah M, Sutamihardja A, Fahle GA, Lyke KE, Laurens MB, Roederer M, Tewari K, Epstein JE, Sim BK, Ledgerwood JE, Graham BS, Hoffman SL; VRC 312 Study Team. Protection against malaria by intravenous immunization with a nonreplicating sporozoite vaccine. Science. 2013 Sep 20;341(6152):1359-65. doi: 10.1126/science.1241800. Epub 2013 Aug 8. PMID 23929949